CLINICAL TRIAL: NCT00357786
Title: An Open-Label Maintenance Study of the Enzyme Replacement Therapy Replagal® (Registered Trademark) in Patients With Fabry Disease
Brief Title: An Open-Label Maintenance Study of the Enzyme Replacement Therapy Replagal in Patients With Fabry Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Raphael Schiffmann, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040027; 04-N-0027
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2008-12

CONDITIONS: Fabry Disease
Keywords: Lysosomal Disease; Glycolipid; Stroke; Peripheral Neuropathy; Storage Disorder
MeSH Terms: conditions — Fabry Disease; Stroke; Peripheral Nervous System Diseases | interventions — agalsidase alfa

ARMS (1):
- A (Experimental): Enzyme replacement for Fabry's Disease
  Interventions: Drug: Replagal agalsidase alfa; Drug: Replagal

INTERVENTIONS:
Drug: Replagal agalsidase alfa
Drug: Replagal

SUMMARY:
This study will continue to evaluate the safety of using intravenous doses of Replagal for two patients with Fabry disease. Fabry disease is a genetic disorder inherited as an X-linked recessive trait. It causes a deficiency in the enzyme alpha galactosidase, which normally breaks down a lipid, or fatty substance called ceramidetrihexoside, a building block in all cells of the body. The deficiency in breaking down the lipid eventually causes that lipid to accumulate and injure cells. Vascular, renal, and neurological problems are the results. It is not known exactly how lipid accumulation brings about such problems, studies of another lipid storage disorder.

Two patients 7 to 17 years of age who have Fabry disease and have been receiving intravenous infusions of Replagal at a dose of 0.2 mg/kg of body weight every 2 weeks may be eligible for this study.

Participants will undergo the following tests and procedures:

* Physical examination.
* Neurological examination.
* Medical and medication history.
* Vital signs.
* Assessment of height and weight.
* Blood tests to determine complete blood count and chemistries.
* Electrocardiogram.
* Doppler blood flow study.

Participants will go through a baseline evaluation, over a period of about 1 day. They will receive an intravenous infusion of Replagal every other week, at the dose of 0.2 mg/kg of body weight. Vital signs will be measured before the infusion and immediately and after and 1 hour afterward. There will be careful monitoring for allergic reactions and side effects. The infusion time takes approximately 40 minutes.

This study will last at least 1 year, or until the sponsor doing the investigating or the drug manufacturer decides to withdraw support of the study.

DETAILED DESCRIPTION:
Objectives: This goal of this study is to continue treating two patients with Fabry disease using enzyme replacement therapy (ERT) using Replagal (agalsidase alfa) at a dose of 0.2 mg/kg of body weight administered every 2 weeks. Study Population: Two patients with Fabry disease who are currently on clinical research protocols 00-N-0185/TKT011 or 02-N-0220/TKT015 and who are stable on ERT. Design: This is an open label study. Outcome Measures: Mainly safety parameters will be obtained. Study duration is estimated to be 2 years.

ELIGIBILITY:
* Patients are under direct care of PI and have previously been treated with Replagal under TKT, Inc. sponsored study numbers 02-N-0220/TKT/010/015.

Ages: 39 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3
Dates: Start 2003-10; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Kidney function | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brady RO, Gal AE, Bradley RM, Martensson E, Warshaw AL, Laster L. Enzymatic defect in Fabry's disease. Ceramidetrihexosidase deficiency. N Engl J Med. 1967 May 25;276(21):1163-7. doi: 10.1056/NEJM196705252762101. No abstract available. PMID 6023233
- [Background] Kahn P. Anderson-Fabry disease: a histopathological study of three cases with observations on the mechanism of production of pain. J Neurol Neurosurg Psychiatry. 1973 Dec;36(6):1053-62. doi: 10.1136/jnnp.36.6.1053. PMID 4204059
- [Background] Kaye EM, Kolodny EH, Logigian EL, Ullman MD. Nervous system involvement in Fabry's disease: clinicopathological and biochemical correlation. Ann Neurol. 1988 May;23(5):505-9. doi: 10.1002/ana.410230513. PMID 3133979